CLINICAL TRIAL: NCT03925922
Title: Comparison Between Fetal Fibronectin (Ffn) vs Cervical Length in Patient With Unfavourable Cervix in Prediction of Successful Induction of Labor
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hytham elhamy, Principal investigator, Ain Shams University
Other Study IDs: Ffn and induction of labour
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Fetal Fibronectin (Ffn)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess the efficacy of fFN compared to transvaginal ultrasound of cervix in prediction of successful induction of labor for unfavorable cervix (bishop score 5 or less).

DETAILED DESCRIPTION:
Induction of labor should be undertaken when the benefits of delivery to either mother or fetus outweigh the risks of pregnancy continuation. Many accepted medical and obstetric indications for labor induction like Hypertensive disorders, Preeclampsia/ eclampsia, Gestational hypertension, Maternal medical conditions, Diabetes mellitus, Renal disease, Chronic pulmonary disease, Chorioamnionitis and Oligohydramnios .Sonographic assessment of cervical length for predicting the outcome of labor induction has been evaluated in numerous studies. The role of ultrasound examination as a tool for selecting women likely to have a successful induction is uncertain . transvaginal sonographic measurements of cervical length in nulliparous women independently predict the likelihood of progress in nulliparous women undergoing labor induction. These observations strongly support the notion that in nulliparous women undergoing labor induction preinduction cervical length plays a key role in labor progression during the latent phase, but not during the active phase of labor .Entering the active phase within 24 hr of induction. On the other hand, cervical length appears to poorly predict the likelihood of cesarean delivery for failure to Bishop's score has the advantage of being universally known . The cutoff point at which delivery can be induced without increasing the risk of cesarean delivery is generally 7 or 6, but this varies from one country to another depending on different local guidelines 6 7 8. However, that point is rarely reached in reality. What's more, Bishop's score does not include parity, even though this variable is known for being closely associated with the induction success. Last, several authors have shown that some components of Bishop's score have a low prognostic value for the success or the failure of the induction .The Bishop score is a poor predictor for the outcome of induced labor at term and should not be used to decide whether to induce labor or not .Fibronectin is large glycoprotein (molecular mass about 420kDa) is normally present in essentially all tissues and body fluids. Its primary function is its role in cell adhesion and phagocytosis .Fetal fibronectin, a glycoprotein thought to act as an adherent at the maternal fetal interface, is uncommonly present in cervicovaginal secretions in the late second and early third trimesters. Although the risk for preterm birth increases as the level of fetal fibronectin rises, it has been evaluated only as a qualitative test, with a value of 50ng/dL or greater being called positive. A positive test is believed to indicate disruption of the maternal-fetal decidual attachment. Asymptomatic women with a positive fetal fibronectin test have an increased risk for preterm birth before 35 weeks, especially within 2 weeks of a positive result. Although the sensitivity of the fibronectin test at 22 to 24 weeks for all spontaneous births before 35 weeks was only 25%, sensitivity for births before 28 weeks was 65% in one study .fFN has been proposed as a new tool for cervical evaluation before labor induction. fFN in cervicovaginal secretion of term deliveries yield a high probability of success of induction women with fibronective negative cervicovaginal secretion and unfavorable cervix score induction of labour should not be attempted .

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous singleton pregnancy
* gestational age between 37week and 42 weeks
* Cephalic presentation
* Bishop score of 5 or less
* No clinical evidence of regular contraction

Exclusion Criteria:

* Rupture of membrane
* Vaginal bleeding
* Any contraindication to vaginal delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females in child bearing period
Study Population: patient will be recruited in this study from those attending to obstetric ER of Ainshams OB/GYN hospital who are nullipara pregnant women gestational age between 37-42 weeks
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Efficacy of fetal fibronectin in prediction of successful induction of labour | 24 hours of induction.
  Comparison between fetal fibronectin versus transvaginal sonography in prediction of successful induction of labour of unfavorable cervix

CONTACTS AND LOCATIONS:
Locations (1):
- AinshamsU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes